CLINICAL TRIAL: NCT04361669
Title: Assessing the Impact of Pharmacist Interventions on Hospice Quality Scores
Brief Title: Hospice Quality Score Assessment Post Pharmacist Intervention
Status: Withdrawn | Type: Observational
Why Stopped: Change in study personnel and sponsor.
Sponsor: Tabula Rasa HealthCare (Industry)
Responsible Party: Sponsor
Other Study IDs: TRHC_RD_Hospice_2020
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Respiratory Disease; Cardiovascular Diseases; Neurologic Disorder; Dementia; Cancer
Keywords: National Quality Forum Score; HCAHPS; Medication refill; Number medications
MeSH Terms: conditions — Respiration Disorders; Cardiovascular Diseases; Nervous System Diseases; Dementia; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: Patients that receive pharmacist-delivered services in the pilot program
  Interventions: Other: Medication safety review
- Control: Patients that do not receive pharmacist-delivered services in the pilot program
  Interventions: Other: Medication safety review

INTERVENTIONS:
Other: Medication safety review — Implementation of a medication safety review using a clinical decision support system

SUMMARY:
The study aims to investigate the impact of pharmacist delivered interventions on hospice patients quality metric scores.

DETAILED DESCRIPTION:
The objective of this study is evaluate a program at a hospice involving activities designed to improve the site's National Quality Forum (NQF) and Consumer Assessment of Healthcare Providers and Systems (HCAHPS) scores. These scores are calculated by the hospice using existing patient satisfaction survey scores (HCAHPS). The institution quantifies their compliance with national quality metrics (NQF) and reports this existing data to the pharmacist providing counseling services to their patients. The pharmacist assesses for areas for improvement and provides additional counseling services to improve the continuity and quality of care. The pilot program is scheduled to launch April 2020 and the researchers will look to assess for changes in the NQF scores, HCAHPS scores, and time for their partnering pharmacy to refill the first set of prescriptions.

ELIGIBILITY:
Inclusion Criteria:

Adult patients who were referred to hospice by a healthcare provider

Exclusion Criteria:

Patients 89 years or older

Ages: 18 Years to 88 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population will be hospice population who received services for 6-months (e.g., between April 2020 to October 2020) and information including: age (excluding patients 89 years or older), gender, medication risk score, NQF score, HCAHPS score, time to fill medication order set, type of chronic condition, and number of medications will be studied.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
National Quality Forum Score | 6 months
  Performance metric used by hospice. Scale 0 - 100 (0=min; 100-high)
Consumer Assessment of Healthcare Providers and Systems | 6 months
  Performance metric used by hospice (0=min; 100-high)
Time to refill | 6 months
  Time to refill prescription from hospice organization (0=min; 100-high)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bingham, PharmD, Principal Investigator — Tabula Rasa HealthCare
Locations (1):
- Tabula Rasa HealthCare, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No